CLINICAL TRIAL: NCT02386150
Title: Phase 1b Escalating Study to Evaluate the Safety and Immunogenicity of Recombinant Ricin Toxin A-Chain 1-33/44-198 (rRTA 1-33/44-198) Vaccine (RVEc™) Administered Intradermally to Healthy Adults as a 3-Dose Primary Series and Booster
Brief Title: ID Recombinant Ricin Toxin A-Chain Vaccine RVEc™ - 3-Dose Primary Series With Boost
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of funding
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: US Army Medical Research Institute of Infectious Diseases (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-14-05; FY14-09 (Other: USAMRIID, Human Use Committee)
Record Dates: First submitted 2015-02-26; First posted 2015-03-11 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Ricin Poisoning
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: 10 μg (Experimental): 10 μg RVEc is to be administered given in the volar surface of the forearm by ID injection (in alternate arms for each vaccination unless there is a medical reason not to alternate arms) with a needle and syringe (ID adapter may be used) (0.1 mL/dose). There are 4 doses planned for this group: 1 primary dose on Days 0, 28, and 106, and a booster dose on Day 365 (1 year).
  Interventions: Biological: RVEc
- Group 2: 20 μg (Experimental): 20 μg RVEc is to be administered given in the volar surface of the forearm by ID injection (in alternate arms for each vaccination unless there is a medical reason not to alternate arms) with a needle and syringe (ID adapter may be used) (0.1 mL/dose). There are 4 doses planned for this group: 1 primary dose on Days 0, 28, and 106, and a booster dose on Day 365 (1 year).
  Interventions: Biological: RVEc

INTERVENTIONS:
Biological: RVEc — The composition of the final drug product, prior to any dilution, is 0.2 mg recombinant ricin toxin 1-33/44-198 (RVEc) in buffer and 0.2% Alhydrogel® at a final volume of 1 mL per vial
  Other Names: Recombinant ricin toxin A-chain 1-33/44-198 (rRTA 1-33/44-198) vaccine

SUMMARY:
This study seeks to determine the safety and immunogenicity of a series of 3 primary vaccinations and a booster vaccination of Recombinant ricin toxin A-chain 1-33/44-198 (rRTA 1-33/44-198) vaccine (RVEc) at 10 or 20 μg intradermally (ID). This study is evaluating if RVEc will display an acceptable safety profile as determined by adverse event (AE) data and if RVEc will elicit anti-ricin antibody titers and ricin toxin-neutralizing antibodies in vaccine recipients.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must read and sign an approved informed consent.
* Study participants must be at least 18 years old at time of screening and no older than 50 years old at time of first study vaccination.
* Participants must weigh at least 110 pounds at time of screening.
* Participants must be in good health as judged from medical history, physical examination, electrocardiogram, chest x-ray, hematology, clinical chemistries, urinalysis, hepatitis serology, and human immunodeficiency virus (HIV) antibody test and must be medically cleared for participation by an investigator.
* Females of childbearing potential must have a negative pregnancy test on screening and the morning of each vaccination prior to receipt of the vaccine and must agree to use a highly effective method of birth control from screening through 3 months following last study vaccination. A highly effective method of birth control is defined as one with a failure rate of less than 1% per year. Acceptable birth control methods that meet this criterion include hormonal implants and injectables, combined oral contraceptives, intrauterine devices, female sterilization (tubal ligation), sexual abstinence, or a vasectomized partner.
* Female participants must also agree not to breastfeed from screening through 3 months following last study vaccination.
* Study participants must be willing to return for all follow-up visits.
* Study participants must agree to report any adverse events (AE) that may or may not be associated with administration of the investigational product through the duration of study participation.
* Study participants must agree to abstain from excessive exercise (more than the usual routine) and excessive alcohol consumption (exceeds 2 drinks for males or exceeds 1 drink for females daily or binge drinking) for the duration of study participation.

Exclusion Criteria:

* Acute or chronic medical conditions or immunodeficiency from a medical condition or medical treatment, medications, or dietary supplements that, in the investigator's opinion, would impair the subject's ability to respond to vaccination. Use of corticosteroids, other than inhaled or topical corticosteroids or eye drops, will not be permitted.
* Severe hypersensitivity to any vaccine.
* History of asthma, chronic obstructive pulmonary disease, or other current/residual diseases of the lungs.
* Clinically significant abnormal laboratory tests. (Normal reference ranges are determined by the local clinical laboratory.)
* Current smoker, to include use of electronic cigarettes.
* Any known allergies to sodium succinate, Polysorbate 20 (a detergent), Alhydrogel, or kanamycin.
* Receipt of any vaccine or investigational product within 30 days before or after vaccination with RVEc (the only exception is the inactivated influenza vaccine that can be received at least 30 days after RVEc Dose 3 or 4).
* Creatine phosphokinase levels that are consistently elevated more than 2 × normal.
* Previous vaccination with RVEc or any other ricin vaccine candidate by any route.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of vaccinated subjects without adverse events by Day 730 | Day 730
  Adverse events will be evaluated for subjects in the assessment population on vaccination days and at follow-up time points.
Percentage of vaccinated subjects with adverse events by Day 730 | Day 730
  Adverse events will be evaluated for subjects in the assessment population on vaccination days and at follow-up time points.
Percentage of vaccinated subjects with any severity of local reactions (Grades 1-4) by Day 730 | Day 730
  Adverse events will be evaluated for subjects in the assessment population on vaccination days and at follow-up time points.
Percentage of vaccinated subjects with system reactions of any severity (Grades 1-4) by Day 730 | Day 730
  Adverse events will be evaluated for subjects in the assessment population on vaccination days and at follow-up time points.
Percentage of vaccinated subjects with generalized allergic reactions by Day 730 | Day 730
  Adverse events will be evaluated for subjects in the assessment population on vaccination days and at follow-up time points.
Percentage of vaccinated subjects with each adverse event by Day 730 | Day 730
  Adverse events will be evaluated for subjects in the assessment population on vaccination days and at follow-up time points.

SECONDARY OUTCOMES:
Total anti-ricin immunoglobulin G (IgG) antibody titers as determined by ELISA | Days 0, 14, 28, 42, 56, 106, 120, 134, 180, 270, 365, 379, 393, 455, 555, 730
Anti-ricin toxin-neutralizing antibody titers as determined by the colorimetric toxin neutralization assay (TNA) | Days 0, 14, 28, 42, 56, 106, 120, 134, 180, 270, 365, 379, 393, 455, 555, 730

CONTACTS AND LOCATIONS:
Overall Officials: Phillip R Pittman, MD, MPH, Principal Investigator — US Army Medical Research Institute of Infectious Diseases
Locations (1):
- Department of Clinical Research, USAMRIID, Fort Deterick, Maryland, United States